CLINICAL TRIAL: NCT02427841
Title: Phase 2 Study of Preoperative Chemotherapy With Abraxane and Gemcitabine Followed by Chemoradiation for Borderline Resectable or Node-Positive Pancreatic Cancer
Brief Title: Nab-paclitaxel and Gemcitabine Hydrochloride Followed by Radiation Therapy Before Surgery in Treating Patients With Pancreatic Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Gina Vaccaro, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011256; NCI-2015-00498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SOL-14124-L; IRB00011256 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2015-04-17; First posted 2015-04-28 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Adenocarcinoma; Resectable Pancreatic Carcinoma
MeSH Terms: interventions — Fluorouracil; dehydroftorafur; Gemcitabine; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, chemoradiation therapy, surgery) (Experimental): PRE-OPERATIVE (NEOADJUVANT) CHEMOTHERAPY: Patients receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-6 weeks after completion of chemotherapy, patients undergo IG-IMRT 5 days a week for 28 fractions and receive fluorouracil IV continuously on days 1-7 for 6 weeks.
  SURGICAL RESECTION: Patients undergo surgery 4-10 weeks after the last dose of chemoradiation.
  POST-OPERATIVE (ADUJUVANT) CHEMOTHERAPY: Beginning within 8-12 weeks after surgery, patients receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4 additional courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Gemcitabine; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine; Gemzar; LY-188011; LY188011
Radiation: Image Guided Radiation Therapy — Undergo IG-IMRT
  Other Names: IGRT; image-guided radiation therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IG-IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; nanoparticle paclitaxel; paclitaxel albumin-stabilized nanoparticle formulation; protein-bound paclitaxel
Procedure: Therapeutic Conventional Surgery — Undergo surgery

SUMMARY:
This phase II trial studies how well nab-paclitaxel and gemcitabine hydrochloride followed by radiation therapy before surgery work in treating patients with pancreatic cancer that can be removed by surgery. Chemotherapy drugs, such as nab-paclitaxel and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving nab-paclitaxel, gemcitabine hydrochloride, and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the R0 (complete resection) resection rate for subjects with borderline resectable or lymph node positive pancreatic adenocarcinoma treated with a multimodality neoadjuvant therapy of preoperative gemcitabine (gemcitabine hydrochloride) and ABRAXANE (nab-paclitaxel) followed by 5-fluorouracil (fluorouracil) based image-guided intensity-modulated radiation therapy (IG-IMRT) chemoradiotherapy.

SECONDARY OBJECTIVES:

I. To determine 1-year relapse-free survival rate with the investigational protocol.

II. To determine 1-year and 2-year overall survival rates. III. To assess response rate by imaging (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) and pathologic analysis.

IV. To assess the toxicity and safety according to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0) criteria.

OUTLINE:

PRE-OPERATIVE (NEOADJUVANT) CHEMOTHERAPY: Patients receive nab-paclitaxel intravenously (IV) over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-6 weeks after completion of chemotherapy, patients undergo IG-IMRT 5 days a week for 28 fractions and receive fluorouracil IV continuously on days 1-7 for 6 weeks.

SURGICAL RESECTION: Patients undergo surgery 4-10 weeks after the last dose of chemoradiation.

POST-OPERATIVE (ADUJUVANT) CHEMOTHERAPY: Beginning within 8-12 weeks after surgery, patients receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4 additional courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed adenocarcinoma of the pancreas
* Tumors must be localized (non-metastatic) and classified as borderline resectable according to Americas Hepato-Pancreato-Biliary Association (AHPBA)/Society of Surgical Oncology (SSO)/Society for Surgery of the Alimentary Tract (SSAT) consensus criteria or be clinically node-positive via computed tomography (CT) or endoscopic ultrasound

  * AHPBA/SSO/SSAT criteria (any one of the following):

    * Tumor-associated deformity of the SMV (superior mesenteric vein) or PV (portal vein)
    * Abutment of the SMV or PV >= 180 degrees
    * Short-segment occlusion of the SMV or PV amenable to resection and venous reconstruction
    * Short-segment involvement of the hepatic artery or its branches amenable to resection and reconstruction
    * Abutment of the superior mesenteric artery (SMA) < 180 degrees
* Subjects must have measurable disease (by RECIST 1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* No prior therapy for pancreatic cancer, including chemotherapy, radiation therapy, definitive surgery or investigational therapy
* Members of all races and ethnic groups will be included
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Absolute neutrophil count >= 1.5 K/cu mm
* Platelets >= 100 K/cu mm
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.25 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance >= 60 mL/min
* No active prior malignancy within 3 years of registration (with the exception of non-melanoma skin cancer, in-situ cancers, or Rai stage 0 chronic lymphocytic leukemia [CLL]); if patient is disease free from a prior malignancy between 3-5 years, special consideration can be requested; in these cases, if the risk of recurrence at 5 years is less than 20%, and in the opinion of the investigator the prior malignancy will not affect the patient's outcome in light of newly diagnosed pancreatic cancer, the patient may be eligible; this will require principle investigator (PI) review and approval on a case by case basis, and approval will be documented in the medical record; all patients who have been disease free from a prior malignancy for at least 5 years will be eligible
* No baseline peripheral sensory neuropathy >= grade 2
* Women of child-bearing potential and men must be willing to use adequate contraception during the entire study and for 8 weeks following completion of all chemotherapy on study; this includes hormonal or barrier method, or abstinence
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Subjects with locally advanced, unresectable primary tumors will not be eligible

  * This includes any of the following:

    * Abutment of the SMA >= 180 degrees
    * Occlusion of the SMV or PV with insufficient normal vein above and below with which to perform venous reconstruction
    * Involvement of the hepatic artery with insufficient artery proximal and distal to perform reconstruction
* Any prior therapy (chemotherapy, radiation or surgery) for pancreatic adenocarcinoma other than biliary decompression
* Subjects who are receiving any other investigational agents
* Subjects with known metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ABRAXANE or other agents used in the study
* Active infection requiring intravenous antibiotics at the time of registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of interstitial lung disease, idiopathic pulmonary fibrosis, silicosis, sarcoidosis or connective tissue disorders (including rheumatoid arthritis and systemic lupus erythematosus)
* Pregnant or breastfeeding women are excluded from this study
* Subjects known to be human immunodeficiency virus (HIV)-positive, including those on combination antiretroviral therapy, are ineligible because of the potential for pharmacokinetic interactions with chemotherapy; in addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy
* Subjects with plastic biliary stents will be excluded; metal biliary stents are allowed and will not be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Vaccaro, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants enrolled who agreed to participate in the study following completion of the informed consent process. 19 started is the number of participants who were assigned to each Arm/Group. One subject withdrew prior to treatment resulting in a total of 19 subjects enrolled and started treatment.
Groups:
- Treatment (Chemotherapy, Chemoradiation Therapy, Surgery): PRE-OPERATIVE (NEOADJUVANT) CHEMOTHERAPY: Patients receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Beginning 3-6 weeks after completion of chemotherapy, patients undergo IG-IMRT 5 days a week for 28 fractions and receive fluorouracil IV continuously on days 1-7 for 6 weeks.
  SURGICAL RESECTION: Patients undergo surgery 4-10 weeks after the last dose of chemoradiation.
  POST-OPERATIVE (ADUJUVANT) CHEMOTHERAPY: Beginning within 8-12 weeks after surgery, patients receive nab-paclitaxel IV over 30 minutes and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 4 additional courses in the absence of disease progression or unacceptable toxicity.
  Fluorouracil: Given IV
  Gemcitabine: Given IV
  Image Guided Radiation Therapy: Undergo IG-IMRT
  Intensity-Modulated Radiation Therapy: Undergo IG-IMRT
  Laboratory Biomarker Analysis: Correlative studies
  Nab-paclitaxel: Given IV
  Therapeutic Conventional Surgery: Undergo surgery
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Started (20 participants enrolled who agreed to participate in the study following completion of the informed consent process. 19 started is the number of participants who were assigned to each Arm/Group. One subject withdrew prior to treatment resulting in a total of 19 subjects enrolled and started treatment.) | 19
Completed | 11
Not Completed | 8
Not completed — Lack of Efficacy | 5
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 68 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) A scale used to describe a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.). Scale ranges from 0 = Fully active, able to carry out all pre-disease performance without restriction to 5 = Dead.
  Participants
    0: Fully Active | 3
    1: Restricted in physically strenuous activity but ambulatory and able to carry out light work | 16
Primary tumor site [Count of Participants; unit: Participants]
  Head | 11
  Body or neck | 5
  Tail | 3
Greatest Tumor diameter [Median (Full Range); unit: cm] | 4.0 [2.0 to 8.9]
Vascular involvement [Count of Participants; unit: Participants]
  Both arterial and venous | 10
  Arterial only | 6
  Venous only | 1
  No vascular involvement | 2
Lymph node status [Count of Participants; unit: Participants]
  Positive nodes on CT scan | 13
  Negative nodes on CT scan | 6
Serum CA 19-9 [Median (Full Range); unit: U/mL] | 231 [4 to 12,414]

OUTCOME MEASURES:

1. Primary Outcome: R0 Resection Rate Defined as Macroscopically Complete Tumor Removal With Negative Microscopic Surgical Margins by Pathologic Assessment
Description: The R0 resection rate, measured as the percent of participants achieving R0 resection among those who initiate study drug, will be computed with 95% confidence interval. A 2-sided binomial test will be used to determine whether the R0 resection rate is significantly greater than 0.37 at 10% significance level.
Time Frame: At the time of surgery
Population: Efficacy evaluable population is those who have received at least one administration of study drug and have at least one efficacy evaluation. Efficacy evaluable participants who fail to go onto surgery are counted as R0 failures (part of the denominator)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
percentage of participants | 42 [20 to 67]
Statistical Analysis 1: Comparison: Treatment (Chemotherapy, Chemoradiation Therapy, Surgery); Study closed early due to lack of enrollment. Study expected to enrolled 44 evaluable patients to achieve 83% power using the 2-sided binomial test at 10% significance. Study enrolled only 19 evaluable patients, meaning the study was underpowered at < 62%; Test type: Superiority — Tested against the standard R0 rate of 37%. Given all evaluable patients are included in the denominator, R0 of 56% was not achieved. Specifically, of the 19 evaluable patients, 11 proceeded to surgery. Of the 11 who underwent surgery, 8 [42% of those enrolled, but 72.7% of those resected] achieved R0 resection; p = .404, 2-sided exact binomial — Study was underpowered; binomial = 42, 95% CI 2-sided [20 to 67] — Test for superiority over standard R0 resection rate of 37%. Study was closed due to slow enrollment, meaning the primary endpoint was underpowered with only 19 of an expected 44 patients enrolled

2. Secondary Outcome: Incidence of Toxicity According to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version (v) 4.0
Description: Frequency and severity of adverse events will be tabulated based on the actual treatment and the number of courses the patient receives. In particular, grade 3 and 4 toxicity rates will be computed and summarized for all patients received at least one dose of the assigned treatment.
Time Frame: From the first dose of study drug(s) until 28 days after last study intervention, up to approximately 3 years, 10 months
Population: Selected adverse reactions with higher incidence (>10%) or notable from package insert (nab-paclitaxel) during pre-operative gemcitabine & nab-paclitaxel therapy per CTCAE terminology version 4.0. N=19
Measure: Number; unit: Adverse Events
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
Adverse Events
  Blood and Lymphatic system disorders | 4
  Gastrointestinal disorders | 24
  Hepatobiliary disorders | 1
  Infections and infestations | 3
  Investigations | 13
  Metabolism and nutrition disorders | 6
  Musculoskeletal and connective tissue disorders | 9
  Nervous system disorders | 15
  Psychiatric disorders | 2
  Respiratory, thoracic and mediastinal disorders | 7
  Skin and subcutaneous tissue disorders | 19
  Vascular disorders | 3

3. Secondary Outcome: Overall Survival Rate Defined as the Percentage of Subjects Alive at the 2 Year Time Point
Description: The expected 2-year overall survival rate (%) will be reported with an associated 95% confidence interval for all enrolled participants (n = 19). Survival is assessed from the first dose of study drug(s) until the date of death due to any cause, up to two years. Participants known still alive at two-years will be censored at two years. Any participant lost to follow up during the two-year period will be censored on the last date known alive.
Time Frame: From first dose of study drug until 2 years or time of death by any cause, which ever comes first. Participants are assessed every 3 months after completing study interventions.
Population: All enrolled participants receiving at least one dose of study drug(s)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
percentage of participants | 41 [24 to 71]

4. Secondary Outcome: Overall Survival Rate Defined as the Percentage of Subjects Alive at the One Year Time Point
Description: The expected 1-year overall survival rate (%) will be reported with an associated 95% confidence interval. Survival is assessed from the first dose of study drug(s) until the date of death due to any cause, up to one year. Participants known still alive at one-year will be censored at one year. Any participant lost to follow up during the one-year period will be censored on the last date known alive.
Time Frame: From first dose of study drug until 1 year or time of death by any cause, whichever comes first. Participants are assessed every 3 months after completing study interventions.
Population: All enrolled participants receiving at least one dose of study drug(s)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
percentage of participants | 79 [63 to 100]

5. Secondary Outcome: Relapse-free Survival Rate Defined as the Percentage of Subjects Who Are Without Recurrence or Death at One Year From Surgical Resection of the Primary Tumor
Description: The expected 1-year relapse-free survival rate (%) will be reported with an associated 95% confidence interval for those who undergo resection (n = 11). Resection-free survival is assessed from the time of resection until time of progression or death by any cause, up to one year. Participants known still alive and without progression at one-year post-resection will be censored at one year. Any participant lost to follow up during the one-year post-resection period will be censored on the last disease assessment date. Response is measured per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 using tumor imaging with CT. Changes in the largest diameter of tumor lesions (target lesions) and shortest diameter of malignant lymph nodes are assessed. Progression is at least 20% increase in sum of diameters of target lesions (referencing nadir sum of diameters) and an absolute increase of at least 5 mm. Presence of any new lesion is also considered progression disease.
Time Frame: From time of resection until progression or death by any cause, within 1 year of resection. Participants are assessed by imaging every 3 months after completing study interventions.
Population: Study participants who receive at least one dose of study drug(s) and undergo surgical resection
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Resection: Those who undergo surgical resection
Arm/Group | Resection
Number analyzed (Participants) | 11
percentage of participants | 64 [41 to 99]

6. Secondary Outcome: Response Rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Defined as the Percent of Subjects With Complete or Partial Disease Response as Confirmed Through Tumor Imaging With Computed Tomography (CT)
Description: The objective response rate (percentage of participants having complete response (CR) or partial response (PR)) will be computed with associated 95% confidence interval using the binomial exact method. Response is measured per RECIST 1.1 using tumor imaging with CT. Changes in the largest diameter of tumor lesions (target lesions) and shortest diameter of malignant lymphnodes are assessed. CR is the disappearance of all target lesions; any pathologic lymph nodes must show a reduction in short axis to < 10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions using the baseline sum of diameters of target lesions as the reference level.
Time Frame: From first dose of study drug(s), with assessments at Staging 1 (approximately 2 months) and Staging 2 (approximately 5 months after first dose of study drug(s)).
Population: Efficacy evaluable population, those receiving at least 1 dose of study drug(s) and having at least 1 efficacy evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
Number analyzed (Participants) | 19
percentage of participants | 21 [6 to 46]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at each investigator office visit from start to conclusion of subject's trial period. (up to 5 years). Utilizing NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0).
Description: Regular investigator assessment.
Arm/Group | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery)
All-Cause Mortality (participants affected / at risk) | 13/19
Serious Adverse Events (participants affected / at risk) | 3/19
Other Adverse Events (participants affected / at risk) | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery) (N=19)
Fascial Dehiscene (Surgical and medical procedures) | 1 (1)
Abdominal wall soft tissue infection (Infections and infestations) | 1 (1)
Intractable Nausea, vomiting, abdominal pain (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
GDA Bleed/Cardiac arrest (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Chemoradiation Therapy, Surgery) (N=19)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenic fever (Blood and lymphatic system disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Abdominal/flank pain (Gastrointestinal disorders) | 2 (2)
Oral mucositis (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)
Edema Limbs (General disorders) | 4 (4)
Fever (General disorders) | 4 (4)
Flu-like symptoms (General disorders) | 4 (4)
Chills (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Hot flashes (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Lethargy (General disorders) | 1 (1)
Localize edema (General disorders) | 1 (1)
Generalized muscle weakness (General disorders) | 1 (1)
Sore throat (General disorders) | 1 (1)
Thrush (General disorders) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Neutropenia (Investigations) | 7 (7)
Thrombocytopenia (Investigations) | 4 (4)
Elevated liver function tests (Investigations) | 2 (2)
Leukopenia (Investigations) | 2 (2)
Hypoalbuminemia (Investigations) | 1 (1)
Elevated pancreatic enzyme (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8)
Dysgeusia (Nervous system disorders) | 3 (3)
DIzziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 7 (7)
Acneiform rash (Skin and subcutaneous tissue disorders) | 2 (2)
Palmar-plantar erythrodyesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Vascular access complication (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study closed early due to lack of enrollment. Study was expected to enrolled 44 evaluable patients to achieve 83% power using the 2-sided binomial test at 10% significance. Study enrolled only 19 evaluable patients, meaning the study was underpowered at < 62%. Study completed stage 1 of Simon's 2-stage minimax design and achieved the required goal of 8 R0 resections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02427841/Prot_SAP_000.pdf